CLINICAL TRIAL: NCT07402837
Title: Creating a Flexible Curriculum Tool for Pediatric Palliative Care Rotating Learners
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Nimisha Bajaj, Co-Principal Investigator, Children's National Research Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: STUDY00001648
Record Dates: First submitted 2026-01-26; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Palliative Care Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Standard Education (Active Comparator): This is the standard palliative care education that most of our learners receive.
  Interventions: Behavioral: Standard Palliative Care Education
- Intervention - Education Using Flexible Curriculum Tool (Experimental): This is the education using a new educational tool that tailors resources, guidance, and education to learner objectives, level of training, learning style, and palliative care experience.
  Interventions: Behavioral: Rotation Using Flexible Education Tool

INTERVENTIONS:
Behavioral: Rotation Using Flexible Education Tool — We are developing a flexible education tool that utilizes a palliative care education database of resources to tailor the structure of a learner rotation to their specific needs. At the moment, education is provided in an ad hoc manner, based on the specific learning objectives, bandwidth of preceptors, and personal knowledge base and resource library. The purpose of this intervention is to provide a standardized database of resources that can be pulled from in an automated manner to design a tailored curriculum for each learner based on their personal learning objectives, learning style, year in training, and experience with palliative care.
  Arms: Intervention - Education Using Flexible Curriculum Tool
Behavioral: Standard Palliative Care Education — This is the typical palliative care education that is provided in an ad hoc manner, based on the specific learning objectives, bandwidth of preceptors, and personal knowledge base and resource library.
  Arms: Control - Standard Education

SUMMARY:
The goal of this clinical trial is to learn if a new educational tool can improve the training and educational process for learners who will already be taking part in the palliative care rotation at Children's National Hospital. The main questions it aims to answer are:

* If learners who are trained using the educational tool more frequently answer strongly agree/agree to the question "I achieved the standard objectives of the palliative care rotation"
* If learners who are trained using the educational tool more frequently answer strongly agree/agree to the question "I achieved my specific objectives of the palliative care rotation"

If there is a comparison group: Researchers will compare responses from learners who did and and did not have their rotation guided by the educational tool to see if there are differences.

Participants will engage in their palliative care rotation as they would have otherwise, though those in the intervention group will be provided different resources. They will be asked to provide responses to survey questions on their end-of-rotation evaluation, and some will be invited to participate in a focus group at the end of their rotation.

ELIGIBILITY:
Inclusion Criteria:

* must be an adult, greater than or equal to 18 years old
* must have rotated with the pediatric palliative care team for at least 1/2 day during the study period
* must speak English

Exclusion Criteria:

* there are no exclusion criteria for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Response to the question "I achieved the standard objectives of the palliative care rotation." | Measured on an evaluation survey sent to participants within 2 weeks after the last day of their rotation, response due within 4 weeks after receipt
  Measured using Likert scale with 5 choices

SECONDARY OUTCOMES:
Response to the question "I achieved my specific objectives of the palliative care rotation." | Measured on an evaluation survey sent to participants within 2 weeks after the last day of their rotation, response due within 4 weeks after receipt
  Measured using Likert scale with 5 choices
Response to the question "I was provided with a variety of resources to meet my learning objectives." | Measured on an evaluation survey sent to participants within 2 weeks after the last day of their rotation, response due within 4 weeks after receipt
  Measured using Likert scale with 5 choices
Response to the question "The education I received matched my level of training." | Measured on an evaluation survey sent to participants within 2 weeks after the last day of their rotation, response due within 4 weeks after receipt
  Measured using Likert scale with 5 choices
Response to the question "The education was appropriate to my previous exposure to hospice and palliative medicine." | Measured on an evaluation survey sent to participants within 2 weeks after the last day of their rotation, response due within 4 weeks after receipt
  Measured using Likert scale with 5 choices
Response to the question "The education on this rotation matched my learning style." | Measured on an evaluation survey sent to participants within 2 weeks after the last day of their rotation, response due within 4 weeks after receipt
  Measured using Likert scale with 5 choices
Response to the question "This rotation was valuable." | Measured on an evaluation survey sent to participants within 2 weeks after the last day of their rotation, response due within 4 weeks after receipt
  Measured using Likert scale with 5 choices
Response to the question "The clinical educators promoted an open, respectful, and safe environment for discussion, learning, and improvement." | Measured on an evaluation survey sent to participants within 2 weeks after the last day of their rotation, response due within 4 weeks after receipt
  Measured using Likert scale with 5 choices
Response to the question "I would recommend this rotation to other learners." | Measured on an evaluation survey sent to participants within 2 weeks after the last day of their rotation, response due within 4 weeks after receipt
  Measured using Likert scale with 5 choices

OTHER OUTCOMES:
Learner confidence in meeting each standard rotation objective before and after the rotation | Measured on an evaluation survey sent to participants within 2 weeks after the last day of their rotation, response due within 4 weeks after receipt
  Measured using a Likert scale of 1-5, in the domains of Patient Care, Medical Knowledge, Interpersonal and Communication Skills, Professionalism, Practice-Based Learning and Improvement, and Systems-Based Practice

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens National Hospital, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2026-02-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT07402837/Prot_000.pdf